CLINICAL TRIAL: NCT02975323
Title: Doppler Ultrasound Hepatic Vein Waveform as a Non-invasive Tool in the Assessment of Severity of Portal Hypertension (DPH Trial)
Brief Title: Doppler Ultrasound Hepatic Vein Waveform as a Non-invasive Tool in the Assessment of Severity of Portal Hypertension
Acronym: DPH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Syed Hasnain Ali Shah, Professor, Aga Khan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-2605/R&D/HEC/12
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Portal Hypertension
Keywords: hepatic venous pressure gradient; liver disease; US Doppler waveform; Cirrhosis
MeSH Terms: conditions — Hypertension, Portal; Liver Diseases; Fibrosis | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single (Experimental): To administer Carvedilol 12.5 mg orally and measure Wedge pressure gradient in hepatic veins followed by change in hepatic vein wave form
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Single dose of oral carvedilol 12.5 mg and wait till the time there's 20% reduction in hepatic wedge pressure gradient from the baseline.
  Other Names: carveda

SUMMARY:
Portal hypertension is the result of an increased hepatic vascular resistance and portal inflow. The best established method to assess portal pressures is the determination of wedged hepatic venous pressure gradient (HVPG). Ultrasound Doppler technique is non-invasive in the assessment of portal hypertension as compared with invasive technique of measurement of the hepatic venous pressure gradient (HVPG). Hemodynamic measurements (BP and pulse recording) will be done and then patient will be given tablet Carvedilol 12.5 mg in a single dose and wait till the time that 20% reduction in heart rate from the baseline occurs. Haemodynamic measurements will be repeated to assess the acute response to beta-adrenoreceptor blocker agent. The change in the HWF will be recorded post beta-adrenoreceptor blocker administration.

DETAILED DESCRIPTION:
Ultrasound Doppler technique is non-invasive in the assessment of portal hypertension as compared with invasive technique of measurement of the hepatic venous pressure gradient (HVPG). The Doppler waveform of the hepatic vein in healthy subjects is normally triphasic (two negative waves and one positive wave) because of central venous pressure variations due to the cardiac cycle. The normal triphasic hepatic vein waveform is transformed into a biphasic or monophasic waveform in patients with cirrhosis. A monophasic waveform has been shown to correlate with a high Child-Pugh score and a poor survival rate.

Therefore, Hepatic vein waveform (HVWF) evaluation with Doppler US may be used as a supplemental tool to assess the severity of Portal Hypertension and therapeutic response to portal pressure lowering drugs in primary prophylaxis of variceal bleed in patients with large oesophageal varices. There's one study which has looked into the same topic but it has been conducted on alcoholic cirrhotics.

Doppler ultrasound is a non-invasive tool in the measurement of portal pressure in portal hypertensive patients. Hemodynamic measurements (BP and pulse recording) will be done and then patient will be given tablet Carvedilol 12.5 mg in a single dose and wait till the time that 20% reduction in heart rate from the baseline occurs. Haemodynamic measurements will be repeated to assess the acute response to beta-adrenoreceptor blocker agent. The change in the HWF will be recorded post beta-adrenoreceptor blocker administration. This study will be a validation and interventional study. It is an open labeled study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis and large varices (≥ 5mm) on screening endoscopy
* Not known esophageal or gastric variceal bleed

Exclusion Criteria:

* Small esophageal varices (<5 mm in size) on screening endoscopy
* Hemodynamically unstable i.e. Blood pressure of <90mmHg and tachycardia of >100bpm.
* Contraindication to Beta-blockers (Asthma, bradycardia, heart failure, allergy)
* history of Esophageal or gastric variceal bleed in the past
* Hepatocellular carcinoma or other metastatic malignancy.
* Portal vein thrombosis (PVT) or Inferior venacaval (IVC) thrombosis
* Congestive cardiac failure (CCF)
* Renal failure or Hepatorenal syndrome (Creatine of >1.5 mg/dl)
* Previous allergy to IV contrast agent.
* Lactating or Pregnant women

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of Correlation of HWF as detected on doppler ultrasound (tri-, bi,- monophasic pattern) and HVPG (mm Hg) as assessed at hepatic vein catherization in the portal hypertensive patient . | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University,, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No